CLINICAL TRIAL: NCT04084249
Title: Implementing Non-invasive Circulating Tumor DNA Analysis to Optimize the Operative and Postoperative Treatment for Patients With Colorectal Cancer - Intervention Trial 2
Brief Title: ctDNA-guided Surveillance for Stage III CRC, a Randomized Intervention Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Claus Lindbjerg Andersen (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Sponsor-Investigator, Claus Lindbjerg Andersen, Professor, Aarhus University Hospital
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IMPROVE-IT2
Record Dates: First submitted 2019-09-04; First posted 2019-09-10 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Colorectal Cancer; Colo-rectal Cancer; ctDNA; Gastro-Intestinal Disorder; Colorectal Neoplasms; Gastrointestinal Cancer; Gastrointestinal Neoplasms; Digestive System Disease; Digestive System Neoplasm; Colonic Diseases; Colonic Neoplasms; Colonic Cancer; Rectal Diseases; Rectal Neoplasms; Rectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Digestive System Diseases; Gastrointestinal Neoplasms; Digestive System Neoplasms; Colonic Diseases; Rectal Diseases; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ctDNA guided surveillance (Experimental): ctDNA analysis will be performed every 4 months postoperatively (4, 8, 12, 16, 20 and 24). At time of first positive ctDNA, patients undergo a whole-body FDG-PET/CT-scan for radiological assessment and a colonoscopy. If the initial assessment is without evidence of recurrence, patients will be offered high-intensive radiological surveillance with FDG-PET/CT-scans every 3 months, until recurrence detection or 21 months has passed. At baseline and months 12, 18, 24 and 36 patients complete the QoL questionnaires including EORTC QLQ-C30, fear of cancer recurrence inventory (FCRI), and impact of events scale for cancer (IES-C). At every FDG-PET/CT-scans the patients also complete the questionnaire.
  Interventions: Diagnostic Test: ctDNA-analysis; Other: Intensified Follow-up Schedule
- Standard Danish follow-up program (No Intervention): Patients will undergo surveillance according to current Danish Guidelines with CT-scans at months 12 and 36 postoperative and colonoscopy every 5 year until age 75. Longitudinal blood samples will be collected at same time-points as in the experimental group but not analyzed until end of trial. At baseline and months 12, 18, 24 and 36 patients complete the QoL questionnaires including EORTC QLQ-C30, fear of cancer recurrence inventory (FCRI), and impact of events scale for cancer (IES-C).

INTERVENTIONS:
Diagnostic Test: ctDNA-analysis — Minimally-invasive blood-based analysis of circulating tumor DNA (ctDNA).
  Arms: ctDNA guided surveillance
Other: Intensified Follow-up Schedule — PET/CT-scans every 3. month
  Arms: ctDNA guided surveillance

SUMMARY:
IMPROVE-IT2 is a randomized multicenter trial comparing the outcomes of ctDNA guided post-operative surveillance and standard-of-care CT-scan surveillance. The hypothesis of this study is that ctDNA guided post-operative surveillance combining ctDNA and radiological assessments could result in earlier detection of recurrent disease and identify more patients eligible for curative treatment.

ELIGIBILITY:
Inclusion Criteria:

* Colon or rectal cancer, tumor stage III (pT1-4N1-2,cM0) or stage II high-risk (pT4N0,cM0 and pT3N0, cM0 with risk factors)
* Have received curative intend resection and be candidates for adjuvant chemotherapy

Exclusion Criteria:

* Not treated with adjuvant chemotherapy
* Synchronous colorectal and non-colorectal cancer diagnosed per-operative (except skin cancer other than melanoma)
* Other cancers (excluding colorectal cancer or skin cancer other than melanoma) within 3 years from screening
* Patients who are unlikely to comply with the protocol (e.g. uncooperative attitude), inability to return for subsequent visits) and/or otherwise considered by the Investigator to be unlikely to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 359 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
FCI | 5 years
  Fraction of patients with relapse receiving intended curative resection or local treatment aiming at complete tumor destruction as defined at the relevant MDT conference.

SECONDARY OUTCOMES:
TTCR | 3 years
  Time to clinical recurrence
3yr-OS | 3 years
  Overall survival at 3 years
5yr-OS | 5 years
  Overall survival at 5 years
QoL | 3 years
  Quality of Life by use of EORTC QLQ-C30, version 3.0. The QoL outcome measure is differences in QLQ-C30 score at 12, 24 and 36 months between the experimental and control arm.
CE | 5 years
  Cost-effectiveness. QoL/Utility weights for the quality-adjusted life years parameter will be QLU-C10D based on EORTC QLQ-C30.
AR | 3 years
  Adherence rate for patients following ctDNA-guided and standard of care surveillance
TTMR | 2 years
  Time to molecular recurrence
FCRI | 3 years
  Fear of Cancer Recurrence Inventory. The FCRI outcome measure is differences in FCRI at 12, 24 and 36 months between the experimental and control arm.
IES-C | 3 years
  Impact of Events Scale Cancer. The IES-C outcome measure is differences in IES-C at 12, 24 and 36 months between the experimental and control arm.

CONTACTS AND LOCATIONS:
Overall Officials: Claus L Andersen, PhD, Principal Investigator — Department of Molecular Medicin, Aarhus University Hospital
Locations (10):
- Denmark (10):
  - Herlev Hospital, Herlev, Capital Region of Denmark
  - Gødstrup Hospital, Herning, Central Jutland
  - Regional Hospital Horsens, Horsens, Central Jutland
  - Regional Hospital Randers, Randers, Central Jutland
  - Aalborg University Hospital, Aalborg, North Denmark
  - Odense University Hospital, Odense, The Region of Southern Denmark
  - Aarhus University Hospital, Aarhus
  - Bispebjerg Hospital, Copenhagen
  - Zealand University Hospital, Køge
  - Regional Hospital Viborg, Viborg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nors J, Henriksen TV, Gotschalck KA, Juul T, Sogaard J, Iversen LH, Andersen CL. IMPROVE-IT2: implementing noninvasive circulating tumor DNA analysis to optimize the operative and postoperative treatment for patients with colorectal cancer - intervention trial 2. Study protocol. Acta Oncol. 2020 Mar;59(3):336-341. doi: 10.1080/0284186X.2019.1711170. Epub 2020 Jan 10. No abstract available. PMID 31920137
- See also: Statistical Analysis Plan — https://www.medrxiv.org/content/10.1101/2024.06.25.24309390v1

DOCUMENTS (2):
  • Study Protocol (2024-07-03): https://cdn.clinicaltrials.gov/large-docs/49/NCT04084249/Prot_002.pdf
  • Statistical Analysis Plan (2024-06-25): https://cdn.clinicaltrials.gov/large-docs/49/NCT04084249/SAP_001.pdf